CLINICAL TRIAL: NCT01507493
Title: The Impact of SCN9A Gene Polymorphism on Individual Pain Perception in the General Population
Status: Completed | Type: Observational
Sponsor: Xianwei Zhang (Other)
Responsible Party: Sponsor-Investigator, Xianwei Zhang, Clinical Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: SCN9A
Record Dates: First submitted 2012-01-02; First posted 2012-01-11 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Pain; Surgery
Keywords: gene polymorphism; SCN9A; pain perception; postoperative pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Heparin anti-coagulated blood (2 ml) was collected from the central venous during the operation and all blood samples were stored at -80℃. Genomic DNA was extracted from the blood samples using a guanidinium isothiocyanate method.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- mutant alleles: grouped by SCN9A mutant alleles including 3312T, 1719R, 1150W.
- wild-type alleles: grouped by SCN9A wild-type alleles including 3312G, 1719C, 1150R.

SUMMARY:
This study was conducted to explore whether the non-synonymous single-nucleotide polymorphisms in SCN9A gene can predict individual basal pain perception and postoperative pain intensity in the general population undergoing upper abdominal surgery. Methods: Patients receiving elective upper abdominal surgery under general anesthesia were recruited into this study. Genotyping of SCN9A was carried out by direct sequencing. The investigators measured their preoperative pressure pain threshold (PPT) and pressure pain tolerance (PTO). The visual analog scale (VAS) was used for pain evaluation at rest during patient-controlled analgesia (PCA) treatment 0 h, 12 h ,24 h and 48h after operation. And the PCA press frequency and drug consumption were recorded.

DETAILED DESCRIPTION:
Patients with the following diseases were excluded: known history of chronic pain, psychiatric diseases or communication disorders, diabetes mellitus, severe cardiovascular diseases, kidney or liver diseases with poor hepatic function, alcohol or drug abuse, heavy smoker, pregnancy or at the lactation period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-70 years
* Receiving elective upper abdominal surgery
* Anesthesiologists (ASA) physical status I or II
* Received PCA administration
* Agreed to participate the research

Exclusion Criteria:

* History of chronic pain
* Psychiatric diseases
* Diabetes mellitus
* Severe cardiovascular diseases
* Kidney or liver diseases
* Alcohol or drug abuse
* Heavy smoker
* Pregnancy or at lactation period
* Refused PCA administration
* Disagree to participate to the research

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 800 Chinese patients receiving elective upper abdominal surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xianwei, Doctor, Study Director — Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mutant Alleles | Wild-type Alleles
Started | 22 | 178
Completed | 22 | 178
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mutant Alleles | Wild-type Alleles | Total
Number analyzed (Participants) | 22 | 178 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 162 | 184
  >=65 years | 0 | 16 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (9.3) | 55.6 (5.3) | 55.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 101 | 113
  Male | 10 | 77 | 87
Region of Enrollment [Number; unit: participants]
  China | 22 | 178 | 200

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption Dose 48h After Operation.
Time Frame: 48 hours after the operation
Measure: Mean (Standard Deviation); unit: microgramme
Arm/Group | Mutant Alleles | Wild-type Alleles
Number analyzed (Participants) | 22 | 178
microgramme | 37.4 (10.4) | 50.4 (20.4)

2. Secondary Outcome: The Visual Analog Scale 48h After Operation.
Description: The visual analog scale (VAS) is used for pain evaluation at rest during patient-controlled analgesia (PCA) treatment 48h after operation. And the visual analog scale is from 0 to 10 which 0 represent no pain while 10 represent unbearable pain
Time Frame: 48 hours after the operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mutant Alleles | Wild-type Alleles
Number analyzed (Participants) | 22 | 178
units on a scale | 6.9 (2.5) | 5.0 (1.7)

3. Secondary Outcome: Preoperative Pressure Pain Threshold (PPT)
Description: The probe of pressure algometer was positioned perpendicularly to the skin surface of the patient, and the investigator applied continuous pressure at approximately the same rate according to the visual LCD display on the algometer. subjects were asked to say "pain" when they started to feel pain during the stimulation. The value from the LCD was recorded as the pressure pain threshold.
Time Frame: 12 hours before the operation
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Mutant Alleles | Wild-type Alleles
Number analyzed (Participants) | 22 | 178
kg/cm2 | 3.6 (1.0) | 3.7 (1.8)

4. Primary Outcome: PCA Press Frequency 48h After Operation.
Time Frame: 48 hours after the operation
Measure: Mean (Standard Deviation); unit: presses per day
Arm/Group | Mutant Alleles | Wild-type Alleles
Number analyzed (Participants) | 22 | 178
presses per day | 8.8 (5.6) | 19.9 (12.7)

5. Secondary Outcome: Preoperative Pressure Pain Tolerance (PTO)
Description: The probe of pressure algometer was positioned perpendicularly to the skin surface of the patient, and the investigator applied continuous pressure at approximately the same rate according to the visual LCD display on the algometer. subjects were asked to say "ok" when they started to feel the pain became intolerable during the stimulation. The value from the LCD was recorded as the pressure pain tolerance.
Time Frame: 12 hours before the operation
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Mutant Alleles | Wild-type Alleles
Number analyzed (Participants) | 22 | 178
kg/cm2 | 6.6 (3.6) | 6.5 (2.6)

ADVERSE EVENTS:
Arm/Group | Mutant Alleles | Wild-type Alleles
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/178
Other Adverse Events (participants affected / at risk) | 0/22 | 0/178

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes